CLINICAL TRIAL: NCT01354327
Title: Study of the Effects of Limicol (a Food Supplement) on LDL-cholesterol in Moderate Hypercholesterolemia Subjects
Brief Title: Effects of Limicol on LDL-cholesterol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lescuyer Laboratory (Industry)
Collaborators: CIC Hôpital de la Conception - Marseille (Unknown); Aix Marseille Université (Other)
Responsible Party: Peltier, Lescuyer Laboratory
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2008-A01169-46
Record Dates: First submitted 2011-05-13; First posted 2011-05-16 (Estimated); Last update posted 2011-05-16 (Estimated); Status verified 2011-05

CONDITIONS: Hypercholesteremia
Keywords: Delivery of Health Care; Cholesterol; LDL-cholesterol; Coronary artery disease; Red yeast rice; Plants extract; Cholesterol excess
MeSH Terms: conditions — Hypercholesterolemia; Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Limicol (Experimental)
  Interventions: Dietary Supplement: Limicol
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Limicol — 3 tablets / day during 4 months
  Arms: Limicol
Dietary Supplement: Placebo — 3 tablets / day during 4 months
  Arms: Placebo

SUMMARY:
The principal objective of this study is to investigate the effects of a novel food supplement (Limicol) on LDL-cholesterol levels in healthy subjects with moderate hypercholesterolemia.

ELIGIBILITY:
Inclusion Criteria:

* About 18 to 55 years (inclusive)
* Subject has a stable weight for at least three months before the start of the study
* Subject able and willing to comply with the protocol and agreeing to give their consent in writing
* Subject affiliated with a social security scheme
* Subject willing to be included in the national register of volunteers who lend themselves to biomedical research

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2008-12; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in blood LDL-cholesterol levels at 4 months | 4 months

SECONDARY OUTCOMES:
Change from Baseline in blood Vit. C, Vit. E, polyphenols and MDA levels at 4 months | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien Peltier, PhD, Study Director — Lescuyer Laboratory
Locations (1):
- Morange, Marseille, France